CLINICAL TRIAL: NCT03906318
Title: Expanded Access Use of Itacitinib to Treat a Single Patient With Aplastic Anemia
Status: No longer available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-39110-18-05
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Iticitinib

SUMMARY:
Expanded Access Use of Itacitinib to Treat a Single Patient With Aplastic Anemia

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Forbes Satter, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital

REFERENCES:
- [Derived] Rosenberg JM, Peters JM, Hughes T, Lareau CA, Ludwig LS, Massoth LR, Austin-Tse C, Rehm HL, Bryson B, Chen YB, Regev A, Shalek AK, Fortune SM, Sykes DB. JAK inhibition in a patient with a STAT1 gain-of-function variant reveals STAT1 dysregulation as a common feature of aplastic anemia. Med. 2022 Jan 14;3(1):42-57.e5. doi: 10.1016/j.medj.2021.12.003. PMID 35590143